CLINICAL TRIAL: NCT02757768
Title: A Phase 4, Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy, Safety, and Tolerability of Mirabegron in Men With Overactive Bladder (OAB) Symptoms While Taking the Alpha Blocker Tamsulosin Hydrochloride for Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Mirabegron in Men With OAB Symptoms While Taking Tamsulosin Hydrochloride for Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Acronym: PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-MA-1008; 2015-004036-36 (EudraCT Number)
Record Dates: First submitted 2016-04-15; First posted 2016-05-02 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Benign Prostatic Hyperplasia; Overactive Bladder
Keywords: Myrbetriq; Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia; Overactive Bladder; Betmiga; Mirabegron; Tamsulosin Hydrochloride
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms | interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirabegron (Experimental): Participants received initial dose of 25 mg of mirabegron which was increased to 50 mg after 4 weeks. In addition to mirabegron participants received 0.4 mg of oral tamsulosin hydrochloride daily throughout the study.
  Interventions: Drug: Mirabegron; Drug: Tamsulosin Hydrochloride
- Placebo (Placebo Comparator): Participants received matching placebo in addition to oral tamsulosin hydrochloride daily throughout the study.
  Interventions: Drug: Placebo; Drug: Tamsulosin Hydrochloride

INTERVENTIONS:
Drug: Mirabegron — Participants received initial dose of 25 mg of mirabegron (oral tablet) which was increased to 50 mg after 4 weeks.
  Other Names: Myrbetriq; Betmiga; YM178
  Arms: Mirabegron
Drug: Placebo — Participants received initial dose of 25 mg of matching placebo (oral tablet) which was increased to 50 mg after 4 weeks.
  Arms: Placebo
Drug: Tamsulosin Hydrochloride — Participants received once daily treatment with tamsulosin hydrochloride 0.4 mg (oral tablet) throughout the study.
  Other Names: Flomax; Omnic

SUMMARY:
The purpose of the study was to assess the efficacy, safety, and tolerability of mirabegron versus placebo in men with overactive bladder (OAB) symptoms while taking tamsulosin hydrochloride for lower urinary tract symptoms (LUTS) due to Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
At Screening (Visit 1), participants entered into a 4-week open label tamsulosin hydrochloride 0.4 mg QD run-in period prior to being randomized into the 12-week double-blind treatment period (Visit 2). At conclusion of the 4-week tamsulosin hydrochloride run-in period, participants completed a 3-day diary just prior to Baseline (Visit 2). Approximately 7 days prior to Visit 2 participants received a phone call reminding them about the diary and to answer any questions.

If participants met all entry criteria at the end of the tamsulosin hydrochloride run-in period, participants were randomized to 1 of 2 treatment groups (mirabegron or placebo) for 12 weeks of treatment in addition to the continuation of tamsulosin hydrochloride 0.4 mg QD. Those participants randomized to Mirabegron started at 25 mg and increased to 50 mg after 4 weeks. Those participants randomized to placebo started blinded product matched to the mirabegron 25 mg tablet and increased to blinded product matched to 50 mirabegron after 4 weeks. Once a participant increased dose, the participant remained on that dose for the remainder of the study unless for safety reasons was required to discontinue study drug.

A training diary was completed in the first 2 weeks of the tamsulosin hydrochloride run-in period. During this evaluation period at least one telephone contact took place with the participant. Diaries were completed at home, using the electronic patient-reported outcome (ePRO) device, for 3 consecutive days prior to each visit: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4), and Week 12/End of Treatment (Visit 5). Site staff contacted the participant approximately 7 days prior to the scheduled visit to remind the participant to complete the electronic diary, review completion instruction and review changes to concomitant medications and adverse events (if applicable).

Three days before Visits 2 (Baseline), 3 (Week 4), 4 (Week 8), and 5 (Week 12), participants completed a 3-day diary, using the ePRO device in which the participant recorded micturition frequency, urgency (PPIUS), incontinence and volume voided. In addition, the diary captured morning and evening blood pressure and pulse rate measurements via Home Blood Pressure Monitoring (HBPM). At Visit 1, International Prostate Symptom Score (IPSS) was completed. At Visits 2, 3, 4, and 5, participants completed the IPSS, EQ-5D-5L, OAB-q, PPBC, and TS-VAS. Maximum urinary flow (Qmax) was measured at Visit 1 (Screening/tamsulosin hydrochloride run-in) and Visit 5 (Week 12/End of Treatment). Post-void residual volume (PVR) was assessed at Screening/tamsulosin hydrochloride run-in (Visit 1), Baseline (Visit 2) and at Week 4 (Visit 3), Week 8 (Visit 4), and Week 12/End of Treatment (Visit 5). A follow-up phone call (Visit 6) was conducted 4-weeks after End of Treatment (Visit 5). Total study participation was approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria assessed at Visit 1 (Screening):

* Men ≥40 years of age with history of overactive bladder (OAB) symptoms (frequency of ≥8 micturitions per day and urgency episodes of ≥2 per day) while taking tamsulosin hydrochloride for at least 2 months to treat LUTS due to BPH.
* Subject has symptoms of OAB (urinary frequency and urgency with or without incontinence) for ≥3 months prior to Screening.
* Subject has an International Prostate Symptom Score (IPSS) score ≥8.
* Subject has Prostate-Specific Antigen (PSA) <4 ng/mL or ≥4 but < 10 ng/mL with a prostate biopsy that is negative for cancer in the past 2 years.
* Subject is willing and able to complete the 3-day diary (including urine volumes, vital signs measurements), and Quality of Life questionnaires.
* Subject and the subject's spouses/partners who are of childbearing potential must be using a highly effective birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS). Birth control must be practiced from Screening and continue throughout the study and for 30 days after the final study drug administration. In addition, sperm donation will not be allowed throughout the study and for 30 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Inclusion Criteria assessed at Visit 2 (Baseline) based on the 3-day diary:

* Subject continues to meet all inclusion criteria of Visit 1 (Screening).
* Subject must experience an average of 8 or more micturitions per day over the 3-day diary period.
* Subject must experience an average of 2 episodes of urgency per day (grade 3 or 4) over the 3-diary period

Exclusion Criteria assessed at Visit 1 (Screening):

* Subject has post-void residual volume (PVR) >200 mL.
* Subject has maximum urinary flow (Qmax) <5.0 mL/second with a minimum voided volume of 125 mL.
* Subject has hematuria >3 rbc/hpf that has not been fully evaluated.
* Subject has evidence of Urinary Tract Infection (UTI). Urine culture and sensitivity will be performed for positive leukocytes, nitrites, or turbidity and will be confirmed with a culture greater than 100,000 cfu/mL. If a subject has a UTI, at Screening (Visit 1) the subject may be rescreened after successful treatment of the UTI (confirmed by a laboratory result of negative urine culture).
* Subject has neurogenic bladder (spinal cord injury, multiple sclerosis, Parkinson's, etc.).
* Subject has diabetic neuropathy.
* Previous open, robotic or minimally invasive prostate surgery (including transurethral procedures). Planned (scheduled) pelvic or prostate surgery during the study period.
* Planned (scheduled) cataract surgery.
* Subject with significant stress incontinence
* Subject with clinically significant bladder outlet obstruction.
* Subject has an indwelling catheter or practices intermittent self-catheterization.
* Subject has experienced 3 or more episodes of recurrent urinary tract infection within the last 12 months.
* Subject has a symptomatic urinary tract infection, prostatitis, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs (i.e., within the confines of the pelvis including the bladder, prostate and rectum; organs of the lower gastrointestinal tract are not necessarily considered pelvic organs such as the distal ascending colon, the full transverse colon and proximal portion of the descending colon are in the abdomen).
* Subject has received intravesical injection in the past 12 months with botulinum toxin, resiniferatoxin, or capsaicin.
* Subject has ever received electro-stimulation therapy for OAB (e.g. sacral nerve stimulation or Percutaneous Tibial Nerve Stimulation [PTNS]).
* Subject began or has changed a bladder training program or pelvic floor exercises less than 30 days prior to Screening.
* Subject has postural hypotension or syncope or postural orthostatic tachycardia.
* Subject has moderate or severe hepatic impairment defined as Child-Pugh Class B or C.
* Subject has severe renal impairment defined as estimated creatinine clearance less than 29 mL/min/1.73 m2 as determined by hospital laboratory calculation of eGFR. A subject with End Stage Renal Disease (ESRD) or undergoing dialysis is also not a candidate for the study.
* Subject has severe uncontrolled hypertension, which is defined as a sitting systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg.
* Subject has baseline resting pulse rate <60 BPM or >90 BPM.
* Subject has evidence of QT prolongation on Screening (Visit 1) or Baseline (Visit 2) electrocardiogram (ECG) defined as QTcF >450 msec.
* Subject has any clinically significant ECG abnormality.
* Subject has AST or ALT >2x upper limit of normal (ULN), or γ-GT >3x ULN and considered clinically significant.
* Subject has a hypersensitivity to any components of mirabegron, tamsulosin hydrochloride, or any of the inactive ingredients.
* Subject has a history of angioedema.
* Subject has any clinical significant condition which makes the subject unsuitable for study participation.
* Subject has been treated with an experimental device within 28 days or received an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* Subject has a concurrent malignancy or history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Subject has ongoing alcohol and/or drug abuse.
* Subject is using prohibited medications within 30 days prior to Screening (Visit 1) through Follow-Up Phone Call (Visit 6).
* Subject has stopped, started or changed the dose of a restricted medication within the 30 days prior to Screening (Visit 1) through Follow-Up Phone Call (Visit 6)
* Subject has participated in an interventional trial within 30 days prior to Screening (Visit 1).
* Subject is involved in the conduct of the study as an employee of the Astellas group, third party associated with the study, or the study site team.
* Subject has previously received mirabegron in the 6 months prior to Screening (Visit 1).

Exclusion Criteria assessed at Visit 2 (Baseline):

* Subject was non-compliant during the 4-week tamsulosin hydrochloride run-in period, defined as taking less than 80% or greater than 120% of study medication.
* Subject had an average total daily urine volume >3000 mL as recorded in the 3-day diary.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc., Medical Affairs, Americas
Locations (79):
- United States (32):
  - Site US01009, Homewood, Alabama
  - Site US01005, Huntsville, Alabama
  - Site US01012, Anchorage, Alaska
  - Site US01070, Hawaiian Gardens, California
  - Site US01081, Los Angeles, California
  - Site US01021, Murrieta, California
  - Site US01068, San Diego, California
  - Site US01064, Valley Village, California
  - Site US01097, Englewood, Colorado
  - Site US01026, Pompano Beach, Florida
  - Site US01025, St. Petersburg, Florida
  - Site US01027, Wellington, Florida
  - Site US01034, West Des Moines, Iowa
  - Site US01094, Shreveport, Louisiana
  - Site US01041, Baltimore, Maryland
  - Site US01016, Boston, Massachusetts
  - Site US01003, Watertown, Massachusetts
  - Site US01060, Kansas City, Missouri
  - Site US01067, Billings, Montana
  - Site US01061, Omaha, Nebraska
  - Site US01029, Edison, New Jersey
  - Site US01031, Albuquerque, New Mexico
  - Site US01015, Garden City, New York
  - Site US01019, Plainview, New York
  - Site US01069, Cary, North Carolina
  - Site US01079, Maiden, North Carolina
  - Site US01072, Bristol, Tennessee
  - Site US01042, Clarksville, Tennessee
  - Site US01056, Knoxville, Tennessee
  - Site US01075, Knoxville, Tennessee
  - Site US01078, Knoxville, Tennessee
  - Site US01063, Newport News, Virginia
- Canada (8):
  - Site CA15008, Calgary, Alberta
  - Site CA15003, Barrie, Ontario
  - Site CA15001, Brampton, Ontario
  - Site CA15005, Toronto, Ontario
  - Site CA15011, Québec, Quebec
  - Site CA15002, Sherbrooke, Quebec
  - Site CA15009, Sherbrooke, Quebec
  - Site CA15014, Victoriaville, Quebec
- Czechia (5):
  - Site CZ42004, Benešov
  - Site CZ42006, Domažlice
  - Site CZ42005, Prague
  - Site CZ42003, Prague
  - Site CZ42001, Sternberk
- France (2):
  - Site FR33004, Colmar
  - Site FR33002, Pierre-Bénite
- Germany (7):
  - Site DE49002, Duisburg
  - Site DE49003, Eisleben Lutherstadt
  - Site DE49001, Hagenow
  - Site DE49006, Halle
  - Site DE49004, Hamburg
  - Site DE49005, Hettstedt
  - Site DE49007, Sangerhausen
- Italy (8):
  - Site IT39002, Avellino
  - Site IT39003, Catanzaro
  - Site IT39010, Chieti
  - Site IT39004, Florence
  - Site IT39005, Latina
  - Site IT39006, Pisa
  - Site IT39001, Treviglio
  - Site IT39008, Vasto
- Poland (5):
  - Site PL48006, Katowice
  - Site PL48001, Piaseczno
  - Site PL48004, Warsaw
  - Site PL48005, Wroclaw
  - Site PL48007, Wroclaw
- Spain (7):
  - Site ES34007, Barcelona
  - Site ES34009, Lugo
  - Site ES34001, Madrid
  - Site ES34003, Miranda de Ebro
  - Site ES34002, Seville
  - Site ES34006, Valencia
  - Site ES34004, Vigo
- United Kingdom (5):
  - Site GB44005, Bristol
  - Site GB44011, Bristol
  - Site GB44004, Newcastle upon Tyne
  - Site GB44002, Reading
  - Site GB44006, York

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled male participants with overactive bladder (OAB) symptoms who were taking the alpha-blocker tamsulosin for lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH).
Pre-assignment Details: Eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled. Participants entered a 4-week open label tamsulosin hydrochloride 0.4 mg once daily (QD) run-in period prior to being randomized in a 1:1 ratio into the 12-week double-blind treatment period of either mirabegron or placebo once daily.
Period: Overall Study
Arm/Group | Mirabegron | Placebo
Started | 356 | 359
Treated | 352 | 354
Completed | 323 | 331
Not Completed | 33 | 28
Not completed — Randomized Never Received Study Drug | 3 | 4
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Deviation | 2 | 9
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Miscellaneous | 4 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population was the all randomized (RAS), which consisted of participants who received initial does of 25 mg of mirabegron or matching placebo which was increased after 4 weeks to 50 mg
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Placebo | Total
Number analyzed (Participants) | 356 | 359 | 715
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (8.3) | 65 (9.5) | 65 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 356 | 359 | 715
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 339 | 336 | 675
  Unknown or Not Reported | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 332 | 325 | 657
  BLACK OR AFRICAN AMERICAN | 16 | 27 | 43
  ASIAN | 4 | 4 | 8
  OTHER | 2 | 2 | 4
  MISSING/UNKNOWN | 2 | 1 | 3
Geographic Region [Count of Participants; unit: Participants]
  Europe | 257 | 257 | 514
  North America | 99 | 102 | 201
Micturition Episodes per 24 Hours [Mean (Standard Deviation); unit: micturitions in 24 hours (M24MIC)] — Population: This baseline measure is based on the full analysis set (FAS), the FAS was defined as all randomized participants who took at least one dose of double-blind treatment after randomization, reported at least one micturition in the baseline diary and at least one micturition post-baseline.
  micturitions in 24 hours (M24MIC) | 10.7 (2.5) | 10.7 (2.6) | 10.7 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Number of Micturitions Per Day
Description: Participants recorded micturitions in the e-diary during three days. The mean number of micturitions was calculated as the average number of times a participant recorded a micturition per day during the 3-day period. Only voluntary micturitions were counted and the episodes of incontinence were not included.
Time Frame: Baseline and Week 12
Population: The analysis population was the full analysis set (FAS), which consisted of all randomized participants who took at least 1 dose of double-blind study drug, reported at least 1 baseline micturition recorded in the 3-day e-diary and at least 1 postbaseline micturition. Last observation carried forward (LOCF) was used for missing values in the EoT.
Measure: Least Squares Mean (Standard Error); unit: micturitions per day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
micturitions per day | -2.00 (0.13) | -1.62 (0.15)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Placebo vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.039, ANCOVA; Least Squares (LS) Mean of Difference = -0.39, 95% CI 2-sided [-0.76 to -0.02], Standard Error of Mean 0.19

2. Secondary Outcome: Change From Baseline to Week 4, Week 8, and Week 12 in Mean Number of Micturitions Per Day
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS.
Measure: Least Squares Mean (Standard Error); unit: micturitions per day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
micturitions per day
  Week 4: number analyzed (Participants) | 334 | 334
  Week 4 | -1.42 (0.13) | -1.32 (0.13)
  Week 8: number analyzed (Participants) | 328 | 326
  Week 8 | -1.89 (0.13) | -1.38 (0.13)
  Week 12: number analyzed (Participants) | 317 | 319
  Week 12 | -1.95 (0.13) | -1.56 (0.13)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Week 4 Placebo vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.558, ANCOVA; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.46 to 0.25], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; Week 8 Placebo vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.007, ANCOVA; LS Mean of Difference = -0.52, 95% CI 2-sided [-0.89 to -0.14], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; Week 12 Placebo vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.041, ANCOVA; LS Mean of Difference = -0.39, 95% CI 2-sided [-0.76 to -0.02], Standard Error of Mean 0.19

3. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition during 3 days of the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: mL per micturition
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
mL per micturition
  Week 4: number analyzed (Participants) | 334 | 333
  Week 4 | 17.74 (1.98) | 13.87 (1.98)
  Week 8: number analyzed (Participants) | 328 | 325
  Week 8 | 22.56 (2.31) | 16.28 (2.32)
  Week 12: number analyzed (Participants) | 317 | 319
  Week 12 | 26.31 (2.53) | 17.32 (2.52)
  EoT | 25.57 (2.42) | 16.32 (2.42)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.167, ANCOVA; LS Mean of Difference = 3.87, 95% CI 2-sided [-1.63 to 9.37], Standard Error of Mean 2.80
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.056, ANCOVA; LS Mean of Difference = 6.29, 95% CI 2-sided [-0.15 to 12.73], Standard Error of Mean 3.28
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.012, ANCOVA; LS Mean of Difference = 8.99, 95% CI 2-sided [1.97 to 16.01], Standard Error of Mean 3.58
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; EoT Placebo vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.007, ANCOVA; LS Mean of Difference = 9.25, 95% CI 2-sided [2.53 to 15.98], Standard Error of Mean 3.43

4. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Mean Number of Incontinence Episodes Per Day
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated as the average number of times a participant recorded an incontinence episode per day during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the full analysis set - incontinence (FAS-I), which consisted of all randomized participants who took at least 1 dose of double-blind study drug and reported 1 micturition at baseline and postbaseline in the 3-day e-diary. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes per day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 132 | 129
incontinence episodes per day
  Week 4: number analyzed (Participants) | 131 | 129
  Week 4 | -0.97 (0.18) | -0.84 (0.18)
  Week 8: number analyzed (Participants) | 130 | 121
  Week 8 | -1.29 (0.22) | -1.20 (0.23)
  Week 12: number analyzed (Participants) | 125 | 119
  Week 12 | -1.48 (0.22) | -1.23 (0.23)
  EoT | -1.45 (0.21) | -1.15 (0.22)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.747, ANCOVA; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.63 to 0.38], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.393, ANCOVA; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.72 to 0.54], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.672, ANCOVA; LS Mean of Difference = -0.25, 95% CI 2-sided [-0.87 to 0.38], Standard Error of Mean 0.32
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.640, ANCOVA; LS Mean of Difference = -0.30, 95% CI 2-sided [-0.90 to 0.30], Standard Error of Mean 0.31

5. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Mean Number of Urgency Episodes (Grade 3 or 4) Per Day
Description: Urgency was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. An urgency episode was defined as any micturition or incontinence episode with a severity of grade 3 or 4, assessed by participants based on the Patient Perception of Intensity of Urgency Scale (PPIUS), where 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could delay voiding a short while; 3 = Severe urgency, could not delay voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The mean number of urgency episodes (grade 3 and/or 4) per day was calculated as the average number of times a participant recorded an urgency episode (grade 3 and/or 4) with or without incontinence per day during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes per day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
urgency episodes per day
  Week 4: number analyzed (Participants) | 334 | 334
  Week 4 | -1.79 (0.15) | -1.53 (0.15)
  Week 8: number analyzed (Participants) | 328 | 326
  Week 8 | -2.68 (0.17) | -1.97 (0.17)
  Week 12: number analyzed (Participants) | 317 | 319
  Week 12 | -2.86 (0.17) | -2.21 (0.17)
  EoT | -2.90 (0.17) | -2.24 (0.17)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.222, ANCOVA; LS Mean of Difference = -0.26, 95% CI 2-sided [-0.68 to 0.16], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.003, ANCOVA; LS Mean of Difference = -0.71, 95% CI 2-sided [-1.18 to -0.24], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.008, ANCOVA; LS Mean of Difference = -0.65, 95% CI 2-sided [-1.13 to -0.17], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.004, ANCOVA; LS Mean of Difference = -0.67, 95% CI 2-sided [-1.13 to -0.21], Standard Error of Mean 0.23

6. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in International Prostate Symptom Score (IPSS) Total Score
Description: The International Prostate Symptom Score (IPSS) consists of 7 questions concerning urinary symptoms and 1 question concerning quality of life (QoL) with total score and subscores (voiding, storage and QoL). The IPSS total score classification ranges from mild (0 to 7) to moderate (8 to 19) or severe (20 to 35). Higher IPSS scored indicated more severe symptoms.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 335 | 330
  Week 4 | -3.9 (0.3) | -4.0 (0.3)
  Week 8: number analyzed (Participants) | 327 | 331
  Week 8 | -5.0 (0.3) | -5.2 (0.3)
  Week 12: number analyzed (Participants) | 318 | 323
  Week 12 | -5.9 (0.3) | -5.5 (0.3)
  EoT: number analyzed (Participants) | 336 | 335
  EoT | -5.7 (0.3) | -5.6 (0.3)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.723, ANCOVA; LS Mean of Difference = 0.1, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.700, ANCOVA; LS Mean of Difference = 0.2, 95% CI 2-sided [-0.7 to 1.0], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.400, ANCOVA; LS Mean of Difference = -0.4, 95% CI 2-sided [-1.3 to 0.5], Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.812, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-1.0 to 0.8], Standard Error of Mean 0.4

7. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in IPSS Subscale Voiding Score
Description: The International Prostate Symptom Score (IPSS) consists of 7 questions concerning urinary symptoms and 1 question concerning quality of life (QoL) with total score and subscores (voiding, storage and QoL). Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The subscale voiding score is the sum of the responses to 4 voiding symptoms questions (incomplete emptying, intermittency, weak stream, and straining). The lowest and highest possible scores range from 0 to 20 (mildly symptomatic to severely symptomatic). A higher score is indicative of worse condition and a negative change from baseline indicates an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 335 | 330
  Week 4 | -1.7 (0.2) | -2.1 (0.2)
  Week 8: number analyzed (Participants) | 327 | 331
  Week 8 | -2.2 (0.2) | -2.5 (0.2)
  Week 12: number analyzed (Participants) | 318 | 323
  Week 12 | -2.5 (0.2) | -2.5 (0.2)
  EoT: number analyzed (Participants) | 336 | 335
  EoT | -2.5 (0.2) | -2.6 (0.2)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.121, ANCOVA; LS Mean of Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.241, ANCOVA; LS Mean of Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.843, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.679, ANCOVA; LS Mean of Difference = 0.1, 95% CI 2-sided [-0.4 to 0.7], Standard Error of Mean 0.3

8. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12, and EoT in IPSS Subscale Storage Score
Description: The International Prostate Symptom Score (IPSS) consists of 7 questions concerning urinary symptoms and 1 question concerning quality of life (QoL) with total score and subscores (voiding, storage and QoL). Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The subscale storage score is the sum of the responses to 3 storage symptoms questions (frequency, urgency, and nocturia). The lowest and highest possible scores range from 0 to 15 (mildly symptomatic to severely symptomatic). A higher score is indicative of worse condition and a negative change from baseline indicates an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 335 | 330
  Week 4 | -2.2 (0.1) | -1.9 (0.1)
  Week 8: number analyzed (Participants) | 327 | 331
  Week 8 | -2.8 (0.2) | -2.6 (0.1)
  Week 12: number analyzed (Participants) | 318 | 323
  Week 12 | -3.3 (0.2) | -3.0 (0.2)
  EoT: number analyzed (Participants) | 336 | 335
  EoT | -3.3 (0.2) | -3.0 (0.2)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.175, ANCOVA; LS Mean of Difference = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.430, ANCOVA; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.141, ANCOVA; LS Mean of Difference = -0.3, 95% CI 2-sided [-0.8 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.288, ANCOVA; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.2

9. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in IPSS Subscale Quality of Life (QoL) Score
Description: The International Prostate Symptom Score (IPSS) consists of 7 questions concerning urinary symptoms and 1 question concerning quality of life (QoL) with total score and subscores (voiding, storage and QoL). The QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The lowest and highest possible score ranges from 0 to 6 (very pleased to terrible). A higher score is indicative of worse condition and a negative change from baseline indicates an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 335 | 330
  Week 4 | -0.9 (0.1) | -0.7 (0.1)
  Week 8: number analyzed (Participants) | 327 | 331
  Week 8 | -1.3 (0.1) | -1.1 (0.1)
  Week 12: number analyzed (Participants) | 318 | 323
  Week 12 | -1.5 (0.1) | -1.3 (0.1)
  EoT: number analyzed (Participants) | 336 | 335
  EoT | -1.4 (0.1) | -1.3 (0.1)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.128, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.054, ANCOVA; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.079, ANCOVA; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.148, ANCOVA; LS Mean of Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.1

10. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Mean Number of Urgency Incontinence Episodes Per Day
Description: Urgency Incontinence was defined as the complaint of involuntary leakage accompanied by or immediately proceeded by urgency. The mean number of urgency incontinence episodes was calculated as the average number of times a participant recorded an urgency incontinence episode per day during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The analysis population was the FAS-I. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes per day
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 132 | 129
urgency incontinence episodes per day
  Week 4: number analyzed (Participants) | 131 | 129
  Week 4 | -0.97 (0.18) | -0.85 (0.18)
  Week 8: number analyzed (Participants) | 130 | 121
  Week 8 | -1.29 (0.22) | -1.19 (0.23)
  Week 12: number analyzed (Participants) | 125 | 119
  Week 12 | -1.52 (0.22) | -1.24 (0.22)
  EoT | -1.49 (0.21) | -1.16 (0.21)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.660, ANCOVA; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.61 to 0.39], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.767, ANCOVA; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.72 to 0.53], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.372, ANCOVA; LS Mean of Difference = -0.28, 95% CI 2-sided [-0.89 to 0.34], Standard Error of Mean 0.31
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.272, ANCOVA; LS Mean of Difference = -0.33, 95% CI 2-sided [-0.92 to 0.26], Standard Error of Mean 0.30

11. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Symptom Bother Score
Description: Overactive bladder symptoms were assessed using the Symptom Bother Scale of the Overactive Bladder questionnaire (OAB-q). The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion consists of 8 questions, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). Lower scores on OAB-q symptom bother indicate a better response.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | -13.73 (0.91) | -11.98 (0.92)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | -18.72 (1.00) | -14.88 (0.99)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | -20.93 (1.07) | -18.03 (1.06)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | -20.18 (1.04) | -18.07 (1.05)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.179, ANCOVA; LS Mean of Difference = -1.75, 95% CI 2-sided [-4.29 to 0.80], Standard Error of Mean 1.30
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.006, ANCOVA; LS Mean of Difference = -3.84, 95% CI 2-sided [-6.60 to -1.08], Standard Error of Mean 1.41
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.055, ANCOVA; LS Mean of Difference = -2.90, 95% CI 2-sided [-5.86 to 0.06], Standard Error of Mean 1.51
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.154, ANCOVA; LS Mean of Difference = -2.11, 95% CI 2-sided [-5.02 to 0.80], Standard Error of Mean 1.48

12. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Total Health Related Quality of Life (HRQL) Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The total score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A higher score on OAB-q HRQL indicated a better response.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | 9.08 (0.80) | 10.43 (0.80)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | 13.06 (0.85) | 13.53 (0.85)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | 15.90 (0.91) | 15.00 (0.90)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | 15.07 (0.89) | 15.12 (0.89)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.233, ANCOVA; LS Mean of Difference = -1.35, 95% CI 2-sided [-3.57 to 0.87], Standard Error of Mean 1.13
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.698, ANCOVA; LS Mean of Difference = 0.46, 95% CI 2-sided [-1.89 to 2.82], Standard Error of Mean 1.20
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.486, ANCOVA; LS Mean of Difference = 0.89, 95% CI 2-sided [-1.62 to 3.40], Standard Error of Mean 1.28
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.968, ANCOVA; LS Mean of Difference = -0.05, 95% CI 2-sided [-2.52 to 2.42], Standard Error of Mean 1.26

13. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in HRQL Subscale Coping Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQL). The HRQL portion consists of 25 HRQL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. A higher score on OAB-q HRQL indicated a better response. The lowest and highest possible scores for the Coping subscale ranges from 8 to 48. The Coping score was calculated by adding the 8 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | 10.58 (0.96) | 12.47 (0.97)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | 16.01 (1.00) | 15.25 (1.00)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | 18.93 (1.09) | 18.03 (1.08)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | 18.05 (1.07) | 18.02 (1.07)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.165, ANCOVA; LS Mean of Difference = -1.89, 95% CI 2-sided [-4.56 to 0.78], Standard Error of Mean 1.36
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.592, ANCOVA; LS Mean of Difference = 0.76, 95% CI 2-sided [-2.02 to 3.54], Standard Error of Mean 1.41
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.559, ANCOVA; LS Mean of Difference = 0.90, 95% CI 2-sided [-2.12 to 3.92], Standard Error of Mean 1.54
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.985, ANCOVA; LS Mean of Difference = 0.03, 95% CI 2-sided [-2.94 to 3.00], Standard Error of Mean 1.51

14. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in HRQL Subscale Concern Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQL). The HRQL portion consists of 25 HRQL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. A higher score on OAB-q HRQL indicated a better response. The lowest and highest possible scores for the Concern subscale ranges from 7 to 42. The Concern score was calculated by adding the 7 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | 9.06 (0.91) | 10.87 (0.92)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | 13.34 (0.98) | 12.99 (0.98)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | 15.64 (1.00) | 14.47 (1.00)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | 14.81 (0.98) | 14.67 (0.99)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.161, ANCOVA; LS Mean of Difference = -1.82, 95% CI 2-sided [-4.35 to 0.72], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.798, ANCOVA; LS Mean of Difference = 0.35, 95% CI 2-sided [-2.36 to 3.07], Standard Error of Mean 1.38
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.408, ANCOVA; LS Mean of Difference = 1.17, 95% CI 2-sided [-1.61 to 3.95], Standard Error of Mean 1.42
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.919, ANCOVA; LS Mean of Difference = 0.14, 95% CI 2-sided [-2.60 to 2.88], Standard Error of Mean 1.39

15. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in HRQL Subscale Sleep Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQL). The HRQL portion consists of 25 HRQL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. A higher score on OAB-q HRQL indicated a better response. The lowest and highest possible scores for the Sleep subscale ranges from 5 to 30. The Sleep score was calculated by adding the 5 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | 10.43 (1.05) | 10.45 (1.06)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | 15.32 (1.10) | 14.41 (1.09)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | 17.94 (1.15) | 16.41 (1.15)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | 16.87 (1.13) | 16.62 (1.13)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.990, ANCOVA; LS Mean of Difference = -0.02, 95% CI 2-sided [-2.94 to 2.91], Standard Error of Mean 1.49
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.554, ANCOVA; LS Mean of Difference = 0.92, 95% CI 2-sided [-2.12 to 3.96], Standard Error of Mean 1.55
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.348, ANCOVA; LS Mean of Difference = 1.53, 95% CI 2-sided [-1.67 to 4.73], Standard Error of Mean 1.63
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.876, ANCOVA; LS Mean of Difference = 0.25, 95% CI 2-sided [-2.89 to 3.38], Standard Error of Mean 1.60

16. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in HRQL Subscale Social Interaction Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQL). The HRQL portion consists of 25 HRQL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. A higher score on OAB-q HRQL indicated a better response. The lowest and highest possible scores for the Social Interaction subscale ranges from 5 to 30. The Social Interaction score was calculated by adding the 5 response scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | 5.55 (0.74) | 6.65 (0.74)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | 8.03 (0.79) | 8.35 (0.79)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | 9.48 (0.79) | 9.57 (0.79)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | 8.96 (0.77) | 9.67 (0.78)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.293, ANCOVA; LS Mean of Difference = -1.10, 95% CI 2-sided [-3.16 to 0.95], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.773, ANCOVA; LS Mean of Difference = -0.32, 95% CI 2-sided [-2.52 to 1.87], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.940, ANCOVA; LS Mean of Difference = -0.08, 95% CI 2-sided [-2.28 to 2.11], Standard Error of Mean 1.12
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.516, ANCOVA; LS Mean of Difference = -0.71, 95% CI 2-sided [-2.86 to 1.44], Standard Error of Mean 1.10

17. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in European Quality of Life in 5 Dimensions and 5 Levels (EQ-5D-5L Questionnaire) Utilities
Description: The EQ-5D-5L is an international standardized non-disease specific generic instrument for describing and valuing health status. It has a multidimensional measure of health-related QoL, capable of being expressed as a single index value and specifically designed to complement other health status measures. The EQ-5D-5L has five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response levels (e.g., 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems/unable to perform the activity). Health-state utility (HSU) data are estimates of the preference for a given state of health on a cardinal numeric scale, where a value of 1.0 represents full health, 0.0 represents dead, and negative values represent states worse than death. Missing EoT values were imputed using LOCF method.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 328 | 320
  Week 4 | 0.011 (0.009) | 0.019 (0.008)
  Week 8: number analyzed (Participants) | 321 | 321
  Week 8 | 0.019 (0.009) | 0.030 (0.009)
  Week 12: number analyzed (Participants) | 313 | 313
  Week 12 | 0.028 (0.009) | 0.032 (0.008)
  EoT: number analyzed (Participants) | 331 | 326
  EoT | 0.026 (0.009) | 0.034 (0.008)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Week 4 Placebo vs. Mirabegron; Test type: Superiority; p = 0.4591, t-test, 2 sided; Statistical comparisons were be made using 2-sided tests at α = 0.05 significance level
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; Week 8 Placebo vs. Mirabegron; Test type: Superiority; p = 0.4073, t-test, 2 sided; Statistical comparisons were be made using 2-sided tests at α = 0.05 significance level
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; Week 12 Placebo vs. Mirabegron; Test type: Superiority; p = 0.7740, t-test, 2 sided; Statistical comparisons were be made using 2-sided tests at α = 0.05 significance level
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; EoT Placebo vs. Mirabegron; Test type: Superiority; p = 0.5121, t-test, 2 sided; Statistical comparisons were be made using 2-sided tests at α = 0.05 significance level

18. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale that asks participants to rate their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems. A higher score indicated a worse perception of bladder condition.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the FAS. Missing values in the EoT were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 330 | 325
  Week 4 | -0.6 (0.1) | -0.5 (0.1)
  Week 8: number analyzed (Participants) | 323 | 325
  Week 8 | -0.8 (0.1) | -0.7 (0.1)
  Week 12: number analyzed (Participants) | 314 | 318
  Week 12 | -1.0 (0.1) | -0.9 (0.1)
  EoT: number analyzed (Participants) | 332 | 330
  EoT | -0.9 (0.1) | -0.9 (0.1)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.223, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.598, ANCOVA; LS Mean of Difference = -0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.312, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.525, ANCOVA; LS Mean of Difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1

19. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Total Urgency and Frequency Score (TUFS)
Description: The TUFS was calculated by adding the PPIUS scores of every void in a participant's 3-day diary, and dividing this by the number of days recorded in the diary. Due to a programming failure in the e-diary data for the number of pads used was not collected.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: The analysis population was the FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale | NA (NA) — Due to a programming failure in the e-diary data for the number of pads used was not collected. | NA (NA) — Due to a programming failure in the e-diary data for the number of pads used was not collected.

20. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Mean Number of Nocturia Episodes Per 24 Hours
Description: A nocturia episode was defined as waking at night one or more time to void (i.e., any voiding associated with sleep disturbance between the date/time the participant goes to bed with the intention to sleep until the date/time the participant gets up in the morning with the intention to stay awake). A night time episode of incontinence is not considered a nocturia episode. The mean number of nocturia episodes per day (24 hours) was calculated as the average number of times a participant recorded a nocturia episode per day during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population was the full analysis set - nocturia (FAS-N), which consisted of all randomized participants who took at least 1 dose of double-blind study drug and reported 1 micturition at baseline and postbaseline in the 3-day e-diary.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes per 24 hours
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 142 | 124
nocturia episodes per 24 hours
  Week 4: number analyzed (Participants) | 141 | 123
  Week 4 | -0.32 (0.07) | -0.45 (0.08)
  Week 8: number analyzed (Participants) | 135 | 118
  Week 8 | -0.48 (0.07) | -0.55 (0.08)
  Week 12: number analyzed (Participants) | 130 | 114
  Week 12 | -0.51 (0.08) | -0.52 (0.08)
  EoT | -0.49 (0.07) | -0.52 (0.08)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.226, ANCOVA; LS Mean of Difference = 0.13, 95% CI 2-sided [-0.08 to 0.34], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.501, ANCOVA; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.14 to 0.28], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.984, ANCOVA; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.22 to 0.23], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.780, ANCOVA; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.18 to 0.24], Standard Error of Mean 0.11

21. Secondary Outcome: Change From Baseline to Week 4, Week 8, Week 12 and EoT in Treatment Satisfaction Visual Analog Scale (TS-VAS)
Description: The TS-VAS is a visual analog scale that asks participants to rate their satisfaction with the treatment by placing a vertical mark on a line that runs from 0 (No, not at all) to 100 (Yes, completely).
Time Frame: Baseline and Weeks 4, 8, and 12
Population: The analysis population consisted of the FAS. LOCF was used for EOT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Mirabegron: Participants received mirabegron at an initial dose of 25 mg, mirabegron was increased to 50 mg after 4 weeks. Participants continued once daily treatment with tamsulosin hydrochloride 0.4 mg throughout the study.
- Placebo: Participants received placebo to match mirabegron at an initial dose of 25 mg, placebo to match mirabegron was increased to 50 mg after 4 weeks. Participants continued once daily treatment with tamsulosin hydrochloride 0.4 mg throughout the study.
Arm/Group | Mirabegron | Placebo
Number analyzed (Participants) | 337 | 339
units on a scale
  Week 4: number analyzed (Participants) | 328 | 324
  Week 4 | 15.6 (1.3) | 12.5 (1.4)
  Week 8: number analyzed (Participants) | 321 | 325
  Week 8 | 18.6 (1.4) | 16.1 (1.4)
  Week 12: number analyzed (Participants) | 313 | 317
  Week 12 | 19.1 (1.5) | 16.9 (1.5)
  EoT: number analyzed (Participants) | 331 | 330
  EoT | 18.4 (1.5) | 16.9 (1.5)
Statistical Analysis 1: Comparison: Mirabegron vs Placebo; Week 4 Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.107, ANCOVA; LS Mean of Difference = 3.1, 95% CI 2-sided [-0.7 to 6.8], Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: Mirabegron vs Placebo; Week 8 Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.190, ANCOVA; LS Mean of Difference = 2.5, 95% CI 2-sided [-1.3 to 6.3], Standard Error of Mean 1.9
Statistical Analysis 3: Comparison: Mirabegron vs Placebo; Week 12 Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.297, ANCOVA; LS Mean of Difference = 2.2, 95% CI 2-sided [-1.9 to 6.3], Standard Error of Mean 2.1
Statistical Analysis 4: Comparison: Mirabegron vs Placebo; EoT Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, age group (<65, >=65 years) and geographical region as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.493, ANCOVA; LS Mean of Difference = 1.4, 95% CI 2-sided [-2.7 to 5.5], Standard Error of Mean 2.1

ADVERSE EVENTS:
Time Frame: From first double-blind medication intake until 30 days after last double-blind medication intake; 16 weeks
Arm/Group | Mirabegron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/352 | 0/354
Serious Adverse Events (participants affected / at risk) | 10/352 | 8/354
Other Adverse Events (participants affected / at risk) | 12/352 | 19/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=352) | Placebo (N=354)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=352) | Placebo (N=354)
Headache (Nervous system disorders) | 6 (6) | 8 (9)
Hypertension (Vascular disorders) | 6 (6) | 11 (12)

LIMITATIONS AND CAVEATS:
The analysis of the EQ-5D endpoint was completed by an external vendor outside of the main study report. Astellas had previously anticipated to post the results in April 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02757768/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT02757768/SAP_001.pdf